CLINICAL TRIAL: NCT04816838
Title: A Window of Opportunity Study for Investigating Drug Tolerant Persister (DTP) to Neoadjuvant Osimertinib in Resectable Non-small Cell Lung Cancer (NSCLC) Harbouring EGFR Mutations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-1335
Record Dates: First submitted 2021-02-24; First posted 2021-03-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N/A(Single Arm) (Experimental)
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — * Osimertinib 80mg once a day(QD) oral(PO)
  Neoadjuvant Period -If there is no disease progression or unacceptable toxicity, treatment is performed for 2cycles at 1 cycle (28 days) interval
  Adjuvant Period
  - If there is no disease progression of unacceptable toxicity, treatment fis performed for 3years at intervals of 1cycle(28days)

SUMMARY:
Osimertinib is a third-generation EGFR (Epidermal growth factor receptor) TKI(Tyrosine kinase inhibitor) for the management of NSCLC(non-small cell lung cancer) harbouring EGFR(Epidermal growth factor receptor) T790M mutation after acquired resistance to previous first-generation EGFR (Epidermal growth factor receptor) TKI(Tyrosine kinase inhibitor) therapy. Moreover, osimertinib was approved or the treatment of patients with EGFR(Epidermal growth factor receptor) mutant NSCLC (non small cell lung cancer) in the first-line setting based on the clinical trial.

The clinical activity and favorable toxicity profile of osimertinib has led to broadly research into this drug as a strategy to inhibit and prevent drug resistance in EGFR(Epidermal growth factor receptor) mutant NSCLC (non small cell lung cancer). Evidences of benefit from EGFR (Epidermal growth factor receptor) TKI(Tyrosine kinase inhibitor) in EGFR(Epidermal growth factor receptor) mutant NSCLC (non small cell lung cancer) patients have been increasing in early stages as well as in advance stages. Therefore, adjuvant or neo adjuvant EGFR (Epidermal growth factor receptor) TKI(Tyrosine kinase inhibitor) in operable NSCLC(non small cell lung cancer) patients could improve survival in EGFR(Epidermal growth factor receptor) mutant NSCLC (non small cell lung cancer) patients.

Acquired resistance by widespread clinical use has become a hot clinical problem.

A variety of target therapies are being developed to overcome tolerance to osimertinib to improve this outcome.

This is an approach that should improve the molecular and clinical understanding of the drug resistance. Specifically, we want to investigate innate drug resistance and tumor microenvironment to osimertinib by performing single-cell RNA sequencing (scRNA-seq). and single cell research is obviously needed to develop cancer therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older
2. Provision of informed consent prior to any study specific procedures
3. Histologically or cytologically confirmed NSCLC(non small cell lung cancer) , performed on a biopsy
4. Documented activating EGFR mutation (Exon 19 deletion or L858R)
5. Positron emission tomography (PET)-computed tomography (CT) within the last 60 days showing radiographic stage I to IIIa lung cancer (mediastinal staging biopsy is allowed but not required)
6. Brain magnetic resonance imaging (MRI) (or CT if contraindication to MRI) within the last 60 days showing no evidence of metastatic disease
7. Documentation that the patient is a candidate for surgical resection of their lung cancer by certified surgeon
8. Measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
9. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1
10. All toxicity from previous chemotherapy, radiation therapy, or surgical procedures according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 recovered to Grade 1 .
11. Patients may receive supplements to meet this requirement this requirement

    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
    * Bilirubin =< 1.5 x ULN (Patients with documented Gilbert's syndrome and conjugated bilirubin within the normal range may be allowed into the study; in this event, it will be documented that the patient was eligible based on conjugated bilirubin levels)
    * Leukocytes > 3,000/mcL
    * Hemoglobin >= 9 g/dL, with no blood transfusions in the 28 days prior to study entry
    * Absolute neutrophil count > 1,500/mcL
    * Platelets > 100,000/mcL
    * Creatinine =< 1.5 x upper limit of normal (ULN) OR creatinine clearance > 50 mL/min/1.73 m2 for patients with creatinine levels =< 1.5 x upper limit above institutional normal
12. Ability to swallow oral medications
13. Women of childbearing potential (WoCBP) must have a negative serum pregnancy test and agree to use highly effective contraception, during the study and for 2 months following the last dose of osimertinib
14. Women NOT of childbearing potential: women who are permanently or surgically sterilized or postmenopausal

    * Permanent sterilization includes hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy but excludes bilateral tubal occlusion; tubal occlusion is considered a highly effective method of birth control but does not absolutely exclude possibility of pregnancy; (the term occlusion refers to both occluding and ligating techniques that do not physically remove the oviducts)
    * Women who have undergone tubal occlusion should be managed on trials as if they are of WoCBP (e.g. undergo pregnancy testing etc., as required by the study protocol)
15. Women will be considered postmenopausal if they are amenorrhoeic for 12 months without an alternative medical cause; the following age-specific requirements apply:

    * Women under 50 years old will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range
    * Women over 50 years of age will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments
16. Acceptable contraception methods are:

    * Total sexual abstinence (abstinence must be for the total duration of the trial and the follow-up period)
    * Vasectomized sexual partner plus male condom (with participant assurance that partner received post-vasectomy confirmation of azoospermia)
    * Tubal occlusion plus male condom
    * Intra-uterine device - provided coils are copper-banded, plus male condom
    * Intra-uterine system (IUS) levonorgestrel IUS (e.g., Mirena), plus male condom
    * Medroxyprogesterone injections (Depo-Provera) plus male condom
    * Etonogestrel implants (e.g., Implanon, Norplant) plus male condom
    * Normal and low dose combined oral contraceptive pills, plus male condom
    * Norelgestromin / ethinylestradiol transdermal system plus male condom
    * Intravaginal device (e.g., ethinylestradiol and etonogestrel) plus male condom
    * Cerazette (desogestrel) plus male condom (Cerazette is currently the only highly efficacious progesterone based pill) For more information, see Appendix E (Definitions of Women of Fertility and Acceptable Contraception Methods).
17. The following methods are considered not to be highly effective and are therefore not acceptable contraceptive methods: - Triphasic combined oral contraceptives; All progesterone only pills except, Cerazette; All barrier methods, if intended to be used alone; Non-copper containing intra-uterine devices; Fertility awareness methods; Coitus interruptus
18. Men must agree to the use of high-efficiency contraception.

Exclusion Criteria:

1. Leptomeningeal carcinomatosis or other central nervous system (CNS) metastases
2. Stage IIIB, or distant metastases (including malignant pleural effusion) identified on PET-CT scan or biopsy
3. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
4. History of confirmed, corneal ulceration
5. Patients who are known to be serologically positive for human immunodeficiency virus (HIV)
6. Active second malignancy, i.e. patient known to have potentially fatal cancer present for which he/she may be (but not necessarily) currently receiving treatment; patients with a history of malignancy that has been completely treated, with no evidence of that cancer currently, are permitted to enroll in the trial provided all chemotherapy for prior malignancy was completed > 12 months prior and/or bone marrow transplant > 2 years prior
7. Patients who are currently receiving treatment with contraindicated corrected QT interval (QTc) prolonging medications or potent CYP3A4 inducers, if that treatment cannot be either discontinued or switched to a different medication prior to first day of study treatment
8. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block.
   * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN) congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes
9. Inadequate bone marrow reserve or organ function (as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count <1.5 x 109/L;
   * Platelet count <100 x 109/L;
   * Haemoglobin <90 g/L;
   * Alanine aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
   * Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
   * Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinaemia] or liver metastases;
   * Serum creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min [measured or calculated by Cockcroft and Gault equation]-confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
10. Treatment with prohibited medications (concurrent anticancer therapy including chemotherapy, radiation, hormonal treatment [except corticosteroids and megesterolacetate], or immunotherapy) =< 14 days prior to treatment with osimertinib
11. Prior treatment with osimertinib or other drugs that target EGFR mutant non-small cell lung cancer (including erlotinib, afatinib, gefitinib, rocelitinib)
12. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, or known active infection including chronic active hepatitis B, hepatitis C and human immunodeficiency virus (HIV); screening for chronic conditions is not required; patients with chronic hepatitis B virus (HBV) with negative HBV viral load on appropriate antiviral therapy will be permitted, if able to continue appropriate antiviral therapy throughout treatment period
13. Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater.
14. Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 week prior) (Appendix DE). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
15. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment, with the exception of alopecia and grade 2 prior platinum-therapy-related neuropathy.
16. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
17. Active tuberculosis
18. Signs or symptoms of infection within 2 weeks prior to first day of study drug treatment
19. Females who are pregnant or breastfeeding
20. Presence of active gastrointestinal (GI) disease (including GI bleeding or ulceration) or other condition that could affect GI absorption (e.g. malabsorption syndrome, history of biliary tract disease), including refractory nausea or vomiting, or chronic GI disease which may affect absorption or tolerance to oral medications
21. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib
22. Involvement in the planning and/or conduct of the study (applies to both investigator staff and/or staff at the study site)
23. Uncontrolled medical, psychological, familial, sociological, or geographical conditions that interfere with the patient's safety, ability to provide informed consent, or ability to comply with the protocol.
24. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rage (ORR) | until 2 years
  after 8 weeks of osimertinib prior to surgery are complete response and partial response determined by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Pathological response rate | A resected tumor specimen is collected during surgery. (Approximately within 10 weeks after dosing)
  * Pathologic complete response rate (pCR): defined as absence of (0%) viable tumor present histologically in the resected tumor specimen
  * Major pathologic response (MPR): ≤10% residual viable tumor following neoadjuvant therapy
Progression Free Survival (PFS) | until 2 years
  The time from curative surgery (no disease) to recurrence/progression/death and From start of osimertinib to documented radiographic relapse/progression by RECIST 1.1 criteria
Overall survival (OS) | After completion of the clinical treatment, subjects are followed up for 30 days and then observed at 3months intervals for up to 1 year.
Ratio of inability to resection (operational to non-surgical conversion rate) | It is performed at study completion, an average of 4year
  Last Patient Performed at the last visit (LPLV). Record the percentage of patients who were initially evaluated as possible to undergo resection and were unable to receive resection due to treatment-related adverse events (AEs) or disease progression.
Incidence of Adverse Events | It is performed at study completion, an average of 4year
  AE captured by CYCAE 5.0 until after 30days of last administration.
Exploratory analysis (Single cell RNA-seq) | Screening, At operation(after 8week of administration)
  perform the analysis of single cell RNA-seq. to characterize heterogeneous gene expression programs within TME and interrelate their transcriptional, functional and genetic diversity between pre and post immunotherapy
Exploratory analysis (Blood sample : PBMC-peripheral blood mononuclear cells) | until 2 years
  perform NGS using SignateraTM assay to detect mutations in the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Sun min Lim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No